CLINICAL TRIAL: NCT01886469
Title: A Phase II, Two-Stage, Open-Label, Single-Treatment, Adaptive Trial Design Examining the Pharmacokinetic and Pharmacodynamic Effects of up to Three Separate HLD100 Modified Release Formulations of Dextroamphetamine Sulfate in Adolescent (Stage 1) and Pediatric (Stage 2) Patients With Attention-Deficit Hyperactivity Disorder.
Brief Title: A Phase II, Adaptive Trial Design Examining the Pharmacokinetic and Pharmacodynamic Effects of Modified Release Amphetamine (HLD100, Formulations B, C and E)) in Adolescents and Children With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLD100-102; HLD100-102 (Control # 163513) (Other: Health Canada)
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Attention-Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (2):
- Adolescents (12-17yrs) (Experimental)
  Interventions: Drug: HLD100-B; Drug: HLD100-C; Drug: HLD100-E
- Children (6-11 yrs) (Experimental)
  Interventions: Drug: HLD100-B; Drug: HLD100-C; Drug: HLD100-E

INTERVENTIONS:
Drug: HLD100-B — d-amphetamine sulfate capsules, 30 mg, CII (25% SR, 30% pH coat, slow release; formulation B)
Drug: HLD100-C — d-amphetamine sulfate capsules, 30 mg, CII (20% SR, 20% pH coat, fast release; formulation E) - this intervention may be deemed unnecessary based on results from Intervention 1.
Drug: HLD100-E — d-amphetamine sulfate capsules, 30 mg, CII (20% SR, 20% pH coat, medium release; formulation E) - this intervention may be deemed unnecessary based on results from Interventions 1 and 2.

SUMMARY:
The main purpose of this study is to determine the rate and extent of absorption of one or more modified release formulations of amphetamine (HLD100) in both adolescents and children with ADHD.

ELIGIBILITY:
Main Inclusion Criteria

* Male and female adolescents (12-17 years; Stage 1) and children (6-11 years; Stage 2).
* Diagnosis of ADHD and confirmed on Kiddie-Schedule for Affective Disorders and Schizophrenia (K-SADS).
* ADHD symptoms controlled on a stable dose of Vyvanse, Adderall XR and or Dexedrine.
* Provision of informed consent (from parent[s] or legal representative[s]) and assent (from subject) for patients.

Main Exclusion Criteria

* Comorbid psychiatric diagnosis (e.g., psychosis, bipolar disorder).
* History of seizures or current diagnosis or family history of Tourette's disorder.
* Use of prescription drugs (except Vyvanse, Dexedrine or Adderall XR) the 14 days and over-the-counter drugs (except birth control) the 30 days before the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Rate and Extent of absorption of d-amphetamine (AUC0-tz, AUC0-∞, Cmax, Tmax, absorption lag time, λz, and t1/2elim) | 48hrs

SECONDARY OUTCOMES:
Safety (AEs, ECG, laboratory parameters, physical examinations) | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Saskatoon Centre for Patient-Oriented Research, Royal University Hospital, Room 5681, C Wing, Saskatoon, Saskatchewan, Canada